CLINICAL TRIAL: NCT02710422
Title: Miami Membrane for Potency (MMeP) Trial to Assess the Impact of Dehydrated Human Amnion Membrane Allograft Placement During Robotic Radical Prostatectomy on Early Return of Erectile Function
Brief Title: Miami Membrane for Potency (MMEP) Trial
Acronym: MMEP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Accrual and Inadequate Funding
Sponsor: University of Miami (Other)
Collaborators: Vivex Biomedical (Unknown)
Responsible Party: Principal Investigator, Sanoj Punnen, Associate Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20150952
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Amniotic Membrane Placement; Robotic Assisted Radical Prostatectomy; RARP; Human Amniotic Membrane Allograft
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prostate-Specific Antigen; Menogaril

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know their treatment arm assignment until after robotic assisted radical prostatectomy (RARP) surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Amniotic Membrane Placement (Experimental): Participants who receive the human amniotic membrane placement after robotic assisted radical prostatectomy (RARP). Participants will also undergo PSA measurement and complete the EPIC 26 and Sexual History Inventory for Men (SHIM) psychosocial questionnaires at protocol-defined intervals.
  Interventions: Biological: Amniotic Membrane Placement; Behavioral: EPIC 26; Other: PSA Measurement; Behavioral: Sexual History Inventory for Men
- Arm 2 - No Amniotic Membrane Placement (Other): Participants who do not receive human amniotic membrane placement after robotic assisted radical prostatectomy (RARP). Participants will also undergo PSA measurement and complete the EPIC 26 and Sexual History Inventory for Men (SHIM) psychosocial questionnaires at protocol-defined intervals.
  Interventions: Behavioral: EPIC 26; Other: PSA Measurement; Behavioral: Sexual History Inventory for Men

INTERVENTIONS:
Biological: Amniotic Membrane Placement — Amniotic membranes will be placed over the neurovascular bundle after extirpative RARP, and before the urethrovesical anastomosis. The membrane will cut into two longitudinal pieces and it will be placed over each neurovascular bundle separately.
  Other Names: Human Amniotic Membrane Allograft
  Arms: Arm 1 - Amniotic Membrane Placement
Behavioral: EPIC 26 — Participants will receive EPIC 26 psychosocial questionnaire at baseline, and post-RARP at protocol-defined intervals.
  Other Names: Expanded Prostate Cancer Index Composite Short Form
Other: PSA Measurement — Measurement of serum PSA levels every three months (+ 1 month) for first year post surgery, and then annually for 5 years.
  Other Names: PSA Test; Prostate Specific Antigen Measurement
Behavioral: Sexual History Inventory for Men — SHIM psychosocial questionnaire administered at baseline, and post-RARP at protocol-defined intervals.
  Other Names: SHIM

SUMMARY:
The use of dehydrated human amnionic membrane allograft improves erectile function recovery (as measured by (Sexual History Inventory for Men (SHIM) score) at 12 months after robotic assisted radical prostatectomy (RARP) compared to a control group with no allograft.

DETAILED DESCRIPTION:
This is a phase 2 prospective randomized trial investigating the impact of amniotic membrane placement over the neurovascular bundles after bilateral nerve sparing robot assisted radical prostatectomy on potency. The study will have a control arm that will follow standard of care surgery, without placement of any membranes. 70 men will be allocated to each arm.

The research study will involve follow up every 3 months for the first 12 months. After this the investigators will follow patients annually with prostate-specific antigen (PSA) measurements and an assessment of any secondary therapies for 5 years post-surgery.

Randomization of study patients will be done in equal proportion to Arm I (membrane placement) and Arm II (no membrane placement, standard of care surgery) using a permuted block design stratified by baseline SHIM score (<17 vs. >=17), and use of ANY erectile aids (Yes vs. No) in the last 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Men age 40-80 with localized prostate cancer who are undergoing bilateral nerve sparing RARP at the University of Miami

Exclusion Criteria:

* Men with poor urinary control at baseline requiring the use of pads for leakage
* Previous treatment for prostate cancer
* Previous history of pelvic radiation
* Men who are using non-oral erectile aids such as vacuum pump, intra-cavernous injections, MUSE, penile prosthesis.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanoj Punnen, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - Amniotic Membrane Placement: Participants who receive the human amniotic membrane placement after robotic assisted radical prostatectomy (RARP). Participants will also undergo PSA measurement and complete the EPIC 26 and Sexual History Inventory for Men (SHIM) psychosocial questionnaires at protocol-defined intervals.
  Amniotic Membrane Placement: Amniotic membranes will be placed over the neurovascular bundle after extirpative RARP, and before the urethrovesical anastomosis. The membrane will cut into two longitudinal pieces and it will be placed over each neurovascular bundle separately.
  EPIC 26: Participants will receive EPIC 26 psychosocial questionnaire at baseline, and post-RARP at protocol-defined intervals.
  PSA Measurement: Measurement of serum PSA levels every three months (+ 1 month) for first year post surgery, and then annually for 5 years.
  SHIM: Psychosocial questionnaire administered at baseline, and post-RARP at protocol-defined intervals.
- Arm 2 - No Amniotic Membrane Placement: Participants who do not receive human amniotic membrane placement after robotic assisted radical prostatectomy (RARP). Participants will also undergo PSA measurement and complete the EPIC 26 and Sexual History Inventory for Men (SHIM) psychosocial questionnaires at protocol-defined intervals.
  EPIC 26: Participants will receive EPIC 26 psychosocial questionnaire at baseline, and post-RARP at protocol-defined intervals.
  PSA Measurement: Measurement of serum PSA levels every three months (+ 1 month) for first year post surgery, and then annually for 5 years.
  SHIM: Psychosocial questionnaire administered at baseline, and post-RARP at protocol-defined intervals.
Period: Overall Study
Arm/Group | Arm 1 - Amniotic Membrane Placement | Arm 2 - No Amniotic Membrane Placement
Started | 12 | 12
3 Month Visit | 9 | 11
6 Month Visit | 7 | 8
9 Month Visit | 5 | 5
12 Month Visit | 3 | 3
Completed | 3 | 3
Not Completed | 9 | 9
Not completed — Termination of study | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Amniotic Membrane Placement | Arm 2 - No Amniotic Membrane Placement | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.33 (6.95) | 61.25 (3.76) | 60.79 (5.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 9 | 12 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
SHIM Score [Mean (Standard Deviation); unit: points on a scale] — Sexual History Inventory for Men (SHIM) psychosocial questionnaire. The SHIM score measures the severity of the participant's Erectile Dysfunction (ED) in points on a scale as follows:
  * 22 - 25: No significant erectile dysfunction
  * 17 - 21: Mild erectile dysfunction
  * 12 - 16: Mild-to-moderate erectile dysfunction
  * 8 - 11: Moderate erectile dysfunction
  * 5 - 7: Severe erectile dysfunction
  points on a scale | 19.25 (7.12) | 21.25 (4.26) | 20.25 (5.83)
PSA Level [Mean (Standard Deviation); unit: ng/mL] — A measure of the amount of prostate-specific antigen (PSA) in the blood.
  ng/mL | 7.29 (3.06) | 6.76 (2.66) | 7.03 (2.82)

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Average Change in SHIM Score, Between Baseline and 12-Months Post-RARP, of Study Participants in Each Group
Description: The difference in average change in Sexual History Inventory for Men (SHIM) score, between baseline and 12 months post RARP between the membrane and control arms will be assessed as the primary endpoint. The SHIM score is measured in points on a scale: The minimum score is 5 to 7 indicating severe erectile dysfunction (ED), the maximum score is 22 to 25, indicating no ED.
Time Frame: Baseline, 12 Months Post-RARP
Population: Due to early study termination, not all study participants completed scheduled visits.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm 1 - Amniotic Membrane Placement | Arm 2 - No Amniotic Membrane Placement
Number analyzed (Participants) | 3 | 3
scores on a scale | 10 (12.288) | 13.33 (6.429)

2. Secondary Outcome: Proportion of Men in Each Group With Mild Erectile Dysfunction (ED) or Better Post-RARP
Description: Among men with a SHIM greater than or equal to 17 at baseline, the investigators will compare the proportion of men in each group with mild ED or better, defined by a SHIM greater than or equal to 17, at 3, 6, 9 and 12 months post RARP.
Time Frame: Baseline, 3, 6, 9 12 Months Post-RARP
Population: Participants with a SHIM score of greater than or equal to 17 at baseline. Due to early study termination, not all study participants completed scheduled visits.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 - Amniotic Membrane Placement | Arm 2 - No Amniotic Membrane Placement
Number analyzed (Participants) | 9 | 9
percentage of participants
  Mild or Better ED, Baseline | 100 | 100
  Mild or Better ED, 3 months: number analyzed (Participants) | 6 | 8
  Mild or Better ED, 3 months | 0 | 0
  Mild or Better ED, 6 months: number analyzed (Participants) | 4 | 5
  Mild or Better ED, 6 months | 0 | 0
  Mild or Better ED, 9 months: number analyzed (Participants) | 4 | 3
  Mild or Better ED, 9 months | 0 | 0
  Mild or Better ED, 12 months: number analyzed (Participants) | 3 | 2
  Mild or Better ED, 12 months | 66.67 | 0

3. Secondary Outcome: Proportion of Men in Each Group Who Are Able to Achieve An Erection Sufficient for Intercourse More the 50% of the Time Post-RARP.
Description: Among men with a SHIM greater than or equal to 17 at baseline, the investigators will compare the proportion of men in each group who are able to achieve an erection sufficient for intercourse more than 50% of the time at 3, 6, 9 and 12 months post RARP.
Time Frame: Baseline, 3, 6, 9 and 12 months Post-RARP
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 - Amniotic Membrane Placement | Arm 2 - No Amniotic Membrane Placement
Number analyzed (Participants) | 9 | 9
percentage of participants
  3 months: number analyzed (Participants) | 6 | 8
  3 months | 0 | 0
  6 months: number analyzed (Participants) | 4 | 5
  6 months | 0 | 0
  9 months: number analyzed (Participants) | 4 | 3
  9 months | 0 | 0
  12 months: number analyzed (Participants) | 3 | 2
  12 months | 66.67 | 0

4. Secondary Outcome: Proportion of Men Who Require the Use of More Invasive Erectile Aids Post-RARP
Description: Among men with a SHIM greater than or equal to 17 at baseline, the investigators will evaluate the proportion of men who require the use of more invasive erectile aids (intra-cavernosal injection, vacuum pump, or penile prosthesis) at 3, 6, 9, and 12 months post RARP.
Time Frame: 3, 6, 9 and 12 Months Post-RARP
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- Arm 1: Amniotic Membrane Placement: Participants who receive the human amniotic membrane placement after robotic assisted radical prostatectomy (RARP). Participants will also undergo PSA measurement and complete the EPIC 26 and Sexual History Inventory for Men (SHIM) psychosocial questionnaires at protocol-defined intervals.
  Amniotic Membrane Placement: Amniotic membranes will be placed over the neurovascular bundle after extirpative RARP, and before the urethrovesical anastomosis. The membrane will cut into two longitudinal pieces and it will be placed over each neurovascular bundle separately.
  EPIC 26: Participants will receive EPIC 26 psychosocial questionnaire at baseline, and post-RARP at protocol-defined intervals.
  PSA Measurement: Measurement of serum PSA levels every three months (+ 1 month) for first year post surgery, and then annually for 5 years.
  SHIM: Psychosocial questionnaire administered at baseline, and post-RARP at protocol-defined intervals.
- Arm 2: No Amniotic Membrane Placement: Participants who do not receive human amniotic membrane placement after robotic assisted radical prostatectomy (RARP). Participants will also undergo PSA measurement and complete the EPIC 26 and Sexual History Inventory for Men (SHIM) psychosocial questionnaires at protocol-defined intervals.
  EPIC 26: Participants will receive EPIC 26 psychosocial questionnaire at baseline, and post-RARP at protocol-defined intervals.
  PSA Measurement: Measurement of serum PSA levels every three months (+ 1 month) for first year post surgery, and then annually for 5 years.
  SHIM: Psychosocial questionnaire administered at baseline, and post-RARP at protocol-defined intervals.
Arm/Group | Arm 1: Amniotic Membrane Placement | Arm 2: No Amniotic Membrane Placement
Number analyzed (Participants) | 9 | 9
percentage of participants
  3 months Post-RARP: number analyzed (Participants) | 6 | 8
  3 months Post-RARP | 0 | 0
  6 months Post-RARP: number analyzed (Participants) | 4 | 5
  6 months Post-RARP | 0 | 0
  9 months Post-RARP: number analyzed (Participants) | 4 | 3
  9 months Post-RARP | 0 | 33.33
  12 months Post-RARP: number analyzed (Participants) | 3 | 2
  12 months Post-RARP | 66.67 | 100

5. Secondary Outcome: Rates of Urinary Control Experienced by Study Participants
Description: Rates of urinary control as measured by no pads per day at 3, 6, 9, and 12 months,
Time Frame: Baseline, 3, 6, 9, and 12 months Post-RARP
Population: Due to early study termination, not all study participants completed scheduled visits.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Amniotic Membrane Placement | Arm 2 - No Amniotic Membrane Placement
Number analyzed (Participants) | 12 | 12
percentage of participants
  No Pad Usage: Baseline | 100 | 100
  No Pad Usage: 3 months post-RARP: number analyzed (Participants) | 9 | 11
  No Pad Usage: 3 months post-RARP | 22.22 | 27.27
  No Pad Usage: 6 months Post-RARP: number analyzed (Participants) | 7 | 8
  No Pad Usage: 6 months Post-RARP | 42.86 | 50
  No Pad Usage: 9 months Post-RARP: number analyzed (Participants) | 5 | 5
  No Pad Usage: 9 months Post-RARP | 60 | 60
  No Pad Usage: 12 months Post-RARP: number analyzed (Participants) | 3 | 3
  No Pad Usage: 12 months Post-RARP | 100 | 33.33

6. Secondary Outcome: 5-year Rate of Prostate Cancer Recurrence Between Both Study Arms
Description: Rate of prostate cancer recurrence in study participants in both study arms at 5 years post-radical prostatectomy.
Time Frame: 5 years post-RARP
Population: Data were not collected due to early termination of study.
Arm/Group | Arm 1 - Amniotic Membrane Placement | Arm 2 - No Amniotic Membrane Placement
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: Per protocol, non-serious adverse events (AEs) were only monitored, assessed and recorded if they were attributed to the membrane placement during the RARP procedure.
Arm/Group | Arm 1 - Amniotic Membrane Placement | Arm 2 - No Amniotic Membrane Placement
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Due to early study termination, not all study participants completed scheduled visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT02710422/Prot_SAP_000.pdf